CLINICAL TRIAL: NCT00235768
Title: Neurotoxicity of Ecstasy: Causality, Course and Clinical Relevance
Brief Title: The NeXT Study; The Netherlands XTC Toxicity Study
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University of Amsterdam, Bonger Institute of Criminology (Unknown); Erasmus Medical Center (Other)
Other Study IDs: ZonMW 310-00-036
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2005-10-10 (Estimated); Status verified 2004-10

CONDITIONS: Ecstasy (Drug); N-Methyl-3,4-Methylenedioxymethamphetamine; Psychopathology
Keywords: Ecstasy; MDMA; Cognition; Brain function; Neuroimaging

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to investigate the possible neurotoxic effects of the party-drug Ecstasy (MDMA)on brain and brain function in humans. Main research questions concern the causality, course and clinical relevance of the neurotoxicity of ecstasy

DETAILED DESCRIPTION:
The study aims to investigate the causality, course and clinical relevance of the observed neurotoxicity in het human brain among users of the popular recreational drug 3,4-methylenedioxymethamphetamine (MDMA). Studies in animals and non-human primates suggest that MDMA is toxic toward brain serotonin neurons at doses that overlap those used by humans. Much less is known about the effects of this drug on the human brain. Recent studies, however, suggest that MDMA might also be neurotoxic to 5-HT neurons in humans, and that it is associated with functional consequences, such as memory impairment and depression. However, these studies have been retrospective and potentially vulnerable to selection bias and confounding. Clearly, only a prospective study can ascertain that recreational XTC is neurotoxic in humans. However, given the existing data such a study is ethically not acceptable. In the present project, therefore, we have chosen a naturalistic study using a combination of prospective and retrospective approaches: a prospective study among 200 XTC naive subjects with a high-risk profile for first XTC use with a two-year follow up of 50 incident-, and 50 continuously XTC naive subjects, and a retrospective design of 25 subjects with and 25 subjects without prior exposure to XTC selected from a large representative cohort (N=1600) that was prospectively followed from the age of 12. In addition, a cross sectional design is used of 70 subjects with variation in type and amount of drugs used, besides a history of frequent XTC use. Among the 50 incident cases and the sample of 50 continuously XTC-naive subjects in the prospective cohort, indicators of neurotoxicity (SPECT,1H-MRS), markers of neuronal injury (fMRI, Perfusion MRI), and clinical assessments of memory, mood and personality prior to any XTC use will be compared with the same parameters two years later, i.e. after XTC user has taken place in the incident cases. In the retrospective cohort, subjects with lifetime XTC exposure will be compared with XTC naive subjects on the same neurotoxicity, neural injury and psychopathology parameters, controlling for potential confounders that were assessed prior to the first use of XTC. In the cross sectional cohort, all subjects will be assessed on the same neurotoxicity, neural injury and psychopathology parameters, controlling for the confounding effects of the use of other psychoactive drugs besides XTC. The combined results will result in conclusions that can be validly used in prevention messages, clinical decision making and the development op a national XTC policy.

ELIGIBILITY:
Inclusion Criteria:

* between 18 - 35 years of age

Exclusion Criteria:

* severe medical or neuropsychiatric illness
* use of prescribed psychotropic medications such as SSRI's
* use of intravenous drugs
* pregnancy
* contra-indications for MRI investigation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225
Dates: Start 2002-04; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Wim van den Brink, MD PhD, Study Director — University of Amsterdam, Academic Medical Center Amsterdam, Dep of Psychiatry; Nick F Ramsey, PhD, Study Director — University Medical Center Utrecht, Dep of Psychiatry; Dirk J Korf, PhD, Study Director — University of Amsterdam, Bonger Institute for Criminology; Maartje ML de Win, MD, Principal Investigator — University of Amsterdam, Academic Medical Center Amsterdam, Dep of Radiology; Gerry Jager, MSc, Principal Investigator — University Medical Center Utrecht, Dep of Psychiatry; Hylke KE Vervaeke, MSc, Principal Investigator — University of Amsterdam, Bonger Institute of Criminology
Locations (3):
- Netherlands (3):
  - Bonger Institute of Criminology, Amsterdam, North Holland
  - Academic Medical Center Amsterdam, Amsterdam, North Holland
  - University Medical Center Utrecht, Utrecht, Utrecht

REFERENCES:
- [Background] de Win MM, de Jeu RA, de Bruin K, Habraken JB, Reneman L, Booij J, den Heeten GJ. Validity of in vivo [123I]beta-CIT SPECT in detecting MDMA-induced neurotoxicity in rats. Eur Neuropsychopharmacol. 2004 May;14(3):185-9. doi: 10.1016/S0924-977X(03)00101-9. PMID 15056477
- [Background] de Win MM, Reneman L, Reitsma JB, den Heeten GJ, Booij J, van den Brink W. Mood disorders and serotonin transporter density in ecstasy users--the influence of long-term abstention, dose, and gender. Psychopharmacology (Berl). 2004 May;173(3-4):376-82. doi: 10.1007/s00213-003-1723-4. Epub 2004 Jan 15. PMID 14726997
- [Background] Reneman L, Booij J, Majoie CB, Van Den Brink W, Den Heeten GJ. Investigating the potential neurotoxicity of Ecstasy (MDMA): an imaging approach. Hum Psychopharmacol. 2001 Dec;16(8):579-588. doi: 10.1002/hup.347. PMID 12404537
- [Background] Reneman L, Endert E, de Bruin K, Lavalaye J, Feenstra MG, de Wolff FA, Booij J. The acute and chronic effects of MDMA ("ecstasy") on cortical 5-HT2A receptors in rat and human brain. Neuropsychopharmacology. 2002 Mar;26(3):387-96. doi: 10.1016/S0893-133X(01)00366-9. PMID 11850153
- [Background] Reneman L, Booij J, de Bruin K, Reitsma JB, de Wolff FA, Gunning WB, den Heeten GJ, van den Brink W. Effects of dose, sex, and long-term abstention from use on toxic effects of MDMA (ecstasy) on brain serotonin neurons. Lancet. 2001 Dec 1;358(9296):1864-9. doi: 10.1016/S0140-6736(01)06888-X. PMID 11741626
- [Background] Reneman L, Majoie CB, Habraken JB, den Heeten GJ. Effects of ecstasy (MDMA) on the brain in abstinent users: initial observations with diffusion and perfusion MR imaging. Radiology. 2001 Sep;220(3):611-7. doi: 10.1148/radiol.2202001602. PMID 11526257
- [Result] De Win MM, Jager G, Vervaeke HK, Schilt T, Reneman L, Booij J, Verhulst FC, Den Heeten GJ, Ramsey NF, Korf DJ, Van den Brink W. The Netherlands XTC Toxicity (NeXT) study: objectives and methods of a study investigating causality, course, and clinical relevance. Int J Methods Psychiatr Res. 2005;14(4):167-85. doi: 10.1002/mpr.6. PMID 16395871